CLINICAL TRIAL: NCT07134764
Title: Evaluation of the Effectiveness of Virtual Reality as an Adjunct to Standard Care in Managing Perioperative Anxiety and Pain in Patients Undergoing Lower Limb Orthopedic Surgery Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sfax (Other)
Responsible Party: Principal Investigator, Fedi Ben Dhaou, PhD Student, University of Sfax
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMS-24-11-1999-51-24
Record Dates: First submitted 2025-08-07; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Perioperative Anxiety; Perioperative Pain Management; Hemodynamic Stability; Satisfaction; Sedative Consumption; Postoperative Complications
Keywords: Virtual reality; Perioperative anxiety; Perioperative pain; Orthopedic surgery; Spinal anesthesia; Randomized controlled trial; Lower limb surgery; Hemodynamic stability
MeSH Terms: conditions — Personal Satisfaction; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in parallel to one of two groups: the intervention group receiving virtual reality exposure during the perioperative period, or the control group receiving standard care. Each participant remains in their assigned group throughout the study, and outcomes will be compared between the two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): Participants in the experimental group will receive an immersive virtual reality (VR) session as an adjunct to standard perioperative care. A SHINECON VR headset will be used to deliver calming or distraction-based visual and auditory content during the entire duration of the orthopedic surgery under spinal anesthesia. The session aims to reduce anxiety and pain perception, minimize the need for sedatives and analgesics, enhance hemodynamic stability, and improve patient and healthcare team satisfaction.
  Interventions: Device: Virtual reality session
- T group (No Intervention): Participants in the control group will receive standard perioperative care as per institutional protocol during orthopedic surgery under spinal anesthesia. No virtual reality device or additional non-pharmacological intervention will be administered. Anxiety, pain, hemodynamic stability, sedative and analgesic use, and satisfaction will be evaluated and compared to the experimental group.

INTERVENTIONS:
Device: Virtual reality session — Patients included in the intervention group (VR group) participated in a comprehensive virtual reality program designed to reduce perioperative anxiety and pain. Prior to their surgery, they attended an introductory VR session aimed at familiarizing them with the technology and providing a calming, immersive environment to help alleviate preoperative stress. Throughout their surgical journey, these patients continued to receive the usual standard care, which included thorough preoperative consultations with healthcare providers, detailed information about the planned surgical procedure, and the provision of standard postoperative care to support recovery. Additionally, during the surgery itself, patients underwent a VR session delivered via a headset, offering real-time immersive distraction and relaxation to minimize intraoperative anxiety and pain perception.
  Arms: VR group

SUMMARY:
The goal of this clinical trial is to evaluate whether virtual reality (VR) can effectively reduce perioperative anxiety and pain in patients undergoing lower limb orthopedic surgery under spinal anesthesia. The study focuses on adult patients in a surgical setting, with an emphasis on improving intraoperative experience and postoperative outcomes without relying solely on pharmacological interventions.

The main questions it aims to answer are:

* Can VR reduce perioperative anxiety and perceived pain levels?
* Does the use of VR lower the need for sedative and analgesic medications and improve hemodynamic stability and satisfaction?

Researchers will compare a VR intervention group to a standard care group to see if VR leads to reduced anxiety and pain, less medication use, better physiological stability, and improved satisfaction.

Participants will:

* Undergo orthopedic surgery under spinal anesthesia.
* Be randomly assigned to either receive standard perioperative care or standard care plus VR immersion.
* In the VR group, engage in calming, immersive virtual environments during the perioperative period.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the effect of immersive virtual reality (VR) on the management of perioperative anxiety and pain in patients undergoing elective lower limb orthopedic surgery under spinal anesthesia. The use of VR as a non-pharmacological adjunct is a novel and promising approach intended to improve the patient's perioperative experience, optimize physiological responses, and potentially reduce the consumption of sedatives and analgesics.

Participants in the intervention group will wear a VR headset that delivers immersive, calming visual and auditory content designed to promote relaxation and distraction before, during, and after the surgical procedure. The control group will receive standard care without VR. Both groups will receive spinal anesthesia as part of routine clinical practice.

Anxiety and pain will be measured at predefined perioperative time points using validated visual analog scales (VAS) and APAIS scale. Additional data on hemodynamic parameters, sedative and analgesic consumption, intraoperative complications, and postoperative satisfaction (from patients, surgeons, and anesthetists) will be collected to evaluate the overall impact of VR on perioperative care quality and patient outcomes.

This study is being conducted at Habib Bourguiba University Hospital, Sfax, Tunisia, over a 12-month period and represents the first clinical evaluation of virtual reality technology in an anesthesia context at this institution. The findings may contribute to the integration of digital tools into routine perioperative care, especially in low-resource settings, by demonstrating their utility in reducing stress, improving comfort, and supporting enhanced recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* - Inclusion Criteria :
* Age between 19 and 64 years
* American Society of Anesthesiologists (ASA) physical status classification I or II (Annex 1)
* Scheduled for lower limb orthopedic surgery under spinal anesthesia
* Provided informed consent to participate in the study
* Non-Inclusion Criteria :
* Patient refusal to participate in the study
* Contraindications to virtual reality (VR) (Patients with cognitive or psychiatric disorders, Claustrophobia, Uncontrolled epilepsy, Visual and/or auditory impairments preventing the use of VR)
* Contraindications to midazolam: known hypersensitivity to benzodiazepines or any excipient of the product
* Patients currently taking anxiolytic medications
* Contraindications to regional anesthesia (spinal anesthesia), (Coagulation disorders, Shock or uncompensated hypovolemia, Unstable arterial hypertension, Decompensated heart failure, Severe aortic or mitral stenosis, Intracranial hypertension, Infection near the puncture site, Progressive neurological disorders, Allergy to local anesthetics, Technical difficulties in performing spinal anesthesia)

Exclusion Criteria:

* Failure of spinal anesthesia requiring conversion to general anesthesia
* Occurrence of an anesthetic or surgical complication
* Occurrence of an adverse effect related to virtual reality, such as (Dizziness, Ocular or muscular contractions triggered by light stimulation, Signs of discomfort : eye strain, blurred vision, disorientation, imbalance, anxiety attack, headache, nausea, vomiting)

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Impact of Immersive Virtual Reality on Reducing Perioperative Anxiety in Lower Limb Orthopedic Surgery Under Spinal Anesthesia | pre during the intervention and post-intervention
  The inversigator expect that the use of immersive virtual reality (VR) during lower limb orthopedic surgery under spinal anesthesia will: Significantly reduce perioperative anxiety levels compared to standard care

SECONDARY OUTCOMES:
The Effect of Virtual Reality on Perioperative Pain, Sedative Use, and Patient Satisfaction in Orthopedic Surgery Under Spinal Anesthesia | pre during the intervention and post-intervention
  The investigator expect that the use of immersive virtual reality (VR) during lower limb orthopedic surgery under spinal anesthesia will:
  * Lower the intensity of perioperative pain as measured by validated pain scales
  * Decrease the need for sedative and analgesic medications during the perioperative period
  * Contribute to more stable hemodynamic parameters during and after the procedure
  * Increase overall satisfaction among patients, as well as anesthesia and surgical teams

CONTACTS AND LOCATIONS:
Overall Officials: Imen Zouche, Professor in Medicine, Study Director — University of Sfax; Yosra Mejdoub, Professor in Medicine, Study Director — University of Sfax
Locations (1):
- Habib Bourguiba University Hospital, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the investigator Publish the Study Article and When the investigator finish Doctoral Studies
Access Criteria: Researchers who may need this data for future studies